CLINICAL TRIAL: NCT05582824
Title: Lactate Metabolism in Patientens With Hyperlactatemia-associated Metabolic Acidosis
Brief Title: Lactate Metabolism in the Hypoperfused Critically Ill
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LacMeta
Record Dates: First submitted 2022-09-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-09

CONDITIONS: Lactate; Metabolism; Hypoperfusion; Metabolomics; Metabolic Acidosis
Keywords: Lactate; Metabolism; Hypoperfusion; Metabolomics; Metabolic Acidosis
MeSH Terms: conditions — Acidosis | interventions — Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main group: All patients included
  Interventions: Other: Blood and urine test

INTERVENTIONS:
Other: Blood and urine test — Daily blood and urine samples

SUMMARY:
Investigating lactate metabolism in critically ill patients whom are hypoperfused by preforming metabolomics via liquid chromatography-mass spectrometry.

DETAILED DESCRIPTION:
Lactate concentration is well known to be directly correlated with risk of death during admission to intensive care. However, lactate by itself is not considered toxic. The study is observational. The breakdown of lactate is being investigated by collecting blood- and urinsamples from patients with hyperlactatemia as a result of hypoperfusion. Levels of lactate, and known as well as unknown metabolites will be identified and quantified by metabolomics. Metabolomics is performed using a combination of liquid chromatography and mass spectrometry. Data will be analysed via statistical analysis to investigate corelations between lactate, a given metabolite and hard outcome such as mortality. And thereby lay the groundwork for potential further research regarding specific lactate-metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sepsis/septic shock or severe heart failure.
* Clinical and paraclinical signs of hypoperfusion in relation to abovementioned diagnosis.
* Metabolic acidosis with s-lactate equal-to-or-above 4 mmol/l.
* Incapacitated

Exclusion Criteria:

* Only regional hypoperfusion such as a leg.
* Receiving intravenous lactate as part of treatment.
* Going in to dialysis. The exclusion is only during dialysis treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A broad spectrum of patients will make up for the population of the study. These are critically ill adults who are admitted to the intensive care unit of Hvidovre Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Laktate levels in blood | Daily testing. Average time frame for the paticipants are 3 days (ranging from 1-10 days).
  Levels of lactate in the blood in relation to the key metabolites (secondary outcomes). Patients included will be testet daily during admission to intensive care whilst lactate is above 2 mmol/l and one more day while laktat is below.

SECONDARY OUTCOMES:
Metabolomics using High Pressure Liquid Cromotografy (HPLC) and Mass Spectrometry (MS) | Two seperate days. One in december 2022 and one in approximately february 2023 (when all patientens are included and all samples are collected).
  Frozen samples collectet during inclusion of patients are analyzed using HPLC and MS which yields results that can later be examined. These results indicate which metabolites are related to, and derived from, lactate. Analasys of blood and urine samples will be done at two seperate days.
Mortality | Admission time ranges up to 6 months.
  Whether or not the patient survived the illness that coursed the admission to the ICU and hospital.
Pyruvate and hydroxybuterate concentration in blood and urine | Two seperate days. One in december 2022 and one in approximately february 2023 (when all patientens are included and all samples are collected).
  Concentration of pyruvate and hydroxybutyrate from blood- and urinsamples are analysed by assays kits on the same occation as metabolomics (HPLC and MS)
Near-infrared spectroscopy (NIRS) | Daily testing. Average time frame for the paticipants are 3 days (ranging from 1-10 days).
  In this case, NIRS consists of two electrodes placed above the eyebrow and on the shoulder. Near-infrared light is sent out by the electrodes to meassure the collour for the blood. Thereby providing information about the oxygen saturation of haemoglobin within the microcirculation.
Peripheral perfusion index (PPI) | Daily testing. Average time frame for the paticipants are 3 days (ranging from 1-10 days).
  PPI is a small clamp around the finger which, like NIRS, uses lightwaves. It measures the ratio of the pulsing blood to non-pulsing blood flow in your finger and is used to indicate the strength of blood flow to your finger. Thereby estimating the microcirculation of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Capital Region, Denmark